CLINICAL TRIAL: NCT05110053
Title: Spinal Cord sTimulation thEraPy for Parkinson's Disease Patients With Gait Problems
Acronym: STEP-PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STEP-PD-449
Record Dates: First submitted 2021-09-23; First posted 2021-11-05 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2023-05

CONDITIONS: Parkinson Disease; Gait Disorders, Neurologic; Fall Injury
MeSH Terms: conditions — Parkinson Disease; Gait Disorders, Neurologic | interventions — Spinal Cord Stimulation

STUDY DESIGN:
Intervention Model Description: Double blinded, placebo-controlled intervention study with six month voluntary, active extension.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Following surgery with implantation of Spinal cord stimulator (SCS), participants will be randomized to either active or placebo stimulation. The patient will have no knowledge of group, as the stimulation protocol is designed to be subperceptional. Further, the primary investigators and outcome assessors will be blinded to group assignment. Imaging analysis will likewise be blinded to group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active (Active Comparator): All patients will receive surgery with implantation of a SCS device. Patients randomized to the active arm, will receive active stimulation. Blinding will continue for 6 months, followed by a 6 month voluntary open-phase, active extension.
  Interventions: Device: Spinal Cord Stimulation
- Placebo (Placebo Comparator): All patients will receive surgery with implantation of a SCS device. Patients randomized to the placebo-arm of the trial will have the device switched off. Blinding will continue for 6 months, followed by a 6 month voluntary open-phase, active extension.
  Interventions: Device: Spinal Cord Stimulation

INTERVENTIONS:
Device: Spinal Cord Stimulation — Spinal Cord stimulation. Surgery is done in local anaesthesia. A small electrode is placed in the epidural space corresponding approximately at the Th8-Th10 level.
  An impulsegenerator, connected to the electrode, is placed in the subcutaneus fat in the gluteal region.

SUMMARY:
Gait difficulties are common in Parkinson's disease (PD) and cause significant disability. No treatment is available for these symptoms. Spinal Cord Stimulation (SCS) has been found to improve gait, including freezing of gait, in a small number of PD patients. The mechanism of action is unclear and some patients are nonresponders.

With this double-blind placebo-controlled proof of concept and feasibility imaging study, we aim to shed light on the mechanism of action of SCS and collect data to inform development of a scientifically sound clinical trial protocol. We also hope to identify imaging biomarkers at baseline that could be predictive of a favourable or a negative outcome of SCS and improve patient selection. Patients will be assessed with clinical rating scales and gait evaluations at baseline and 6 and 12 months after SCS. They will also receive serial 18F-FDG and ([18F]FEOBV) PET scans to assess the effects of SCS on cortical/subcortical activity and brain cholinergic function

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a chronic neurodegenerative disorder affecting almost 2% of all people over the age of 65 worldwide. Based on records from the nationwide Danish Hospital Register, 1,931 patients with a first-time diagnosis of PD were seen in Danish hospitals between 2001 and 2006, and according to the Danish Parkinson Association, more than 8,000 people live in Denmark with PD, but many more people, including relatives and caregivers, are affected by the burden of the disease. The pathological hallmark of PD is the loss of dopaminergic projection neurons in the substantia nigra, manifesting as the classic triad of bradykinesia, rigidity and tremor. These symptoms can be effectively treated with dopamine replacement therapy, at least in the initial stages of the disease. However, as the disease progresses, more debilitating symptoms occur, including gait problems, postural instability, and falls. Unfortunately, the occurrence of these symptoms represents a major milestone in PD progression, resulting in loss of independence, worsened quality of life, and markedly increased mortality (from the consequences of falls e.g. hip fractures). Average survival is reduced to 7 years once a PD patient starts having falls. The socioeconomic cost of falls in PD is also significant, with 80% of spending on PD care arising from acute admissions, primarily falls related. Gait problems, postural instability, and falls in PD, like in the non-PD elderly population, are multi-factorial. However, there are PD-specific factors that contribute to the onset of these symptoms, including deficits of central sensory processing and motor deficits such as freezing of gait (FoG). Critically, these disabling symptoms often respond poorly to dopaminergic drugs, and advanced therapy, including subthalamic nucleus deep brain stimulation (DBS). Recent work has implicated cholinergic dysfunction in PD secondary to degeneration of brainstem locomotor regions such as the Pedunculopontine nucleus (PPN), which is involved in the control of movement initiation and body equilibrium. However, so far, the response of postural and locomotor symptoms to interventions such as cholinesterase inhibitors or PPN DBS (that both enhance cholinergic neurotransmission) has been disappointing with a great deal of variability in reported responses among patients. This variability in treatment response to therapy is probably related to the heterogeneity of mechanisms of postural and gait abnormalities across the PD population, suggesting the importance of phenotyping PD patients with postural and gait problems when starting a therapeutic agent or recruiting patients in clinical studies to investigate new strategies for these problems.

Spinal cord stimulation (SCS) is an established therapy to treat chronic back and neuropathic pain.

Several studies have shown an improvement in gait function in PD patients following SCS for back pain. More recently, a small number of PD patients with gait dysfunction (without back pain) were treated with encouraging initial results on gait function and with few adverse events. However, the trials performed so far have left a number of unanswered questions with SCS that need to be addressed before this procedure can be used more widely in PD patients with gait problems. Firstly, all the published studies are unblinded and carried out in small cohorts of PD patients. Secondly, while these studies have shown that, overall, SCS seems to have a beneficial effect on gait in PD, they have also shown a heterogeneous outcome, as some patients had a poor response to treatment. Thirdly, patient selection and gait characterisation in these studies was limited, and this lack of clinical phenotyping could have been responsible for the heterogeneous outcome of these studies. Fourthly, mechanisms of actions of SCS are uncertain/unstudied in these papers. Therefore, a prospective, double-blind clinical trial with a scientifically sound study protocol in larger cohort of well-characterised patients is required in order to provide clear Class I evidence whether SCS is effective in improving gait function in PD. Additionally, the exact mechanisms of action of SCS in PD patients with gait problems are uncertain, as they have not been fully investigated so far. Animal models of PD, including non-human primates, show that SCS improves locomotion by activating the dorsal column-medial lemniscal pathway which in turn desynchronizes abnormal corticostriatal oscillations. Inputs from ascending leminiscal and extralemniscal pathways to the brainstem and thalamus that may modulate the supplementary motor area (SMA) are also highly connected to the cholinergic PPN in the brainstem. In turn, the SMA has cortifugal projections to PPN, as part of the circuit that controls anticipatory postural adjustments. Therefore, SCS might modulate the activity of SMA, globus pallidus and PPN that are impaired in patients with FoG.

Positron Emission Tomography (PET) can be used to assess in vivo these changes induced by SCS on the brain cholinergic function and the motor and associative cortical-subcortical loops.

([18F]FEOBV) PET is an in vivo marker of the brain vesicular acetylcholine transporter (VAChT) and provides information of the functional integrity of the brain cholinergic neurotransmitter system. Using ([18F]FEOBV) PET we have recently showed reduced striatal and limbic archicortical VAChT binding in patients who suffer from FoG compared to participants who do not suffer from this. 18F-deoxyglucose (18F-FDG) PET is a marker of regional cerebral glucose metabolic rate (rCMRglc), Over the last three decades, studies of regional cerebral glucose metabolism have provided insight into the pathophysiology of the cerebral dysfunction underlying PD and other movement disorders. 18F-FDG PET has also been extensively used to assess the effects of pallidotomy and DBS on the motor and associative cortical-subcortical loops.

Therefore, PET imaging with ([18F]FEOBV) PET and 18F-FDG before and after SCS treatment could significantly improve the understanding of the mechanisms of actions of SCS and its effects on brain cholinergic neurotransmission and resting metabolic brain networks. This knowledge may be helpful in selecting the right patient group for the procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Idiopathic PD diagnosed by a movement disorders neurologist
2. Presence of gait functional impairment despite optimal medical management
3. Able to walk independently without an aid for a minimum of two minutes without rest
4. Absence of secondary causes of gait problems
5. Able to understand study requirements - able to provide consent
6. Above 50 years of age

Exclusion Criteria:

1. The presence of another significant neurological/psychiatric disorder or significant disease
2. Spinal anatomical abnormalities precluding SCS surgery
3. History of stroke or structural lesions on CT that could interfere with image analysis.
4. History of chronic pain and severe degenerative spine disease with or without chronic pain
5. History of drug addiction or dependency
6. Previous DBS surgery for PD
7. Pregnancy or breast-feeding.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Clinical improvement of gait | Follow-up at 6 and 12 months
  To establish proof of concept by changes in Postural Instability and Gait Difficulty (PIGD) subscore of the Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS UPDRS). This subscore is the sum of 2.12 (Walking and balance), 2.13 (Freezing), 3.10 (Gait), 3.11 (Freezing of gait) and 3.12 (Postural stability)
Changes in resting metabolic networks assessed with 18-FDG PET/CT | Follow-up at 6 and 12 months
  18-FDG is a tracer characterizing glucose metabolism. Quantification of 18F-FDG PET scans will be performed. Analysis of PET scans will be performed using both a region of interest (ROI) approach sampling hypothesized areas and exploratory Statistical Parametric Mapping (SPM). For each subject, ROIs will be defined on the individual CT and copied onto co-registered PET images. ROIs will include putamen, caudate nuclei, ventral striatum, thalamus, red nucleus, amygdala, hypothalamus, locus coeruleus, median raphe and the ventral tegmental area. SPM will allow automated interrogation of parametric images across the whole brain volume at a voxel level to localize significant differences in tracer uptake without a priori selection of target regions.
  The primary end points are the between-group differences in striatal and extrastriatal tracer uptake/binding.
Changes in brain cholinergic function | Follow-up at 6 and 12 months
  ([18F]FEOBV) PET is an in vivo marker of the brain vesicular acetylcholine transporter (VAChT) and provides information of the integrity of the brain cholinergic neurotransmitter system. Quantification of 18FEOBV scans will be performed. Analysis of PET scans will be performed using both a region of interest (ROI) approach sampling hypothesized areas and exploratory Statistical Parametric Mapping (SPM). For each subject, ROIs will be defined on the individual CT and copied onto co-registered PET images. ROIs will include putamen, caudate nuclei, ventral striatum, thalamus, red nucleus, amygdala, hypothalamus, locus coeruleus, median raphe and the ventral tegmental area. SPM will allow automated interrogation of parametric images across the whole brain volume at a voxel level to localize significant differences in tracer uptake without a priori selection of target regions.
  The primary end points are the between-group differences in striatal and extrastriatal tracer uptake/binding.
Adverse events | 6 and 12 months
  Evaluation of the safety and tolerability of SCS treatment in patients with PD. Measured as type, frequency and severity of adverse events.

SECONDARY OUTCOMES:
subjective changes in quality of life per SF-36 | Follow-up at 6 and 12 months
  Subjective changes in symptom severity and improvements in quality of life as measured by Short Form-36
subjective changes in parkinsons specific quality of life | Follow-up at 6 and 12 months
  Subjective changes in symptom severity and improvements in quality of life as measured by Parkinsons Disease Quality of Life questionnaire (PDQ-39)
Clinical improvement of gait as measured by TUG in s | Follow-up at 6 and 12 months
  Objective changes in gait function as assessed by timed up and go test (TUG), measured in seconds
subjective changes in gait function | Follow-up at 6 and 12 months
  Subjective changes in symptom severity and improvements in quality of life as measured by Acitivities-specific Balance Confidence scale (ABC)
subjective changes in occurence of freezing | Follow-up at 6 and 12 months
  Subjective changes in symptom severity and improvements in quality of life as measured by the Freezing of Gait Questionnaire (FOGQ)
Overall Changes in PD severity | Follow-up at 6 and 12 months
  Overall changes in symptoms of PD, assessed by the Movement Disorder Society Unified Parkinsons Disease Rating Scale (MDS-UPDRS)
Improvement in home based gait ability | Follow-up at 6 and 12 months
  Objective changes in gait function at home using biometric data, collected by the patients themselves using a waist-worn triaxial accelerometer
Changes in cognitive function as assessed by moca | Follow-up at 6 and 12 months
  Assessed by MoCA
Clinical improvement of balance as measured by BBS | Follow-up at 6 and 12 months
  Objective changes in gait function as assessed by Berg Balance Scale, scored 0-56, higher scores being better

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Pavese, MD, PhD, FRCP, FEAN, Principal Investigator — University of Aarhus
Locations (1):
- Aarhus University, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Yes
As a significant amount of imaging data will be collected over the course of this trial, this data may be made available upon request based upon the relevance and scientific merit of the request.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Upon request
Access Criteria: Based on relevant request to a principal investigator

REFERENCES:
- [Derived] Terkelsen MH, Hvingelby VS, Johnsen EL, Moller M, Danielsen EH, Henriksen T, Glud AN, Tai Y, Baun AM, Knudsen AL, Valdemarsen RN, Horsager J, Okkels N, Andersen ASM, Meier K, Borghammer P, Molloy S, Nandi D, Moro E, Sorensen JCH, Pavese N. Spinal cord stimulation therapy for gait impairment in Parkinson's disease: a double-blinded, randomised feasibility trial with an open extension. Nat Commun. 2026 Jan 29. doi: 10.1038/s41467-026-68782-w. Online ahead of print. PMID 41611672
- [Derived] Hvingelby VS, Hojholt Terkelsen M, Johnsen EL, Moller M, Danielsen EH, Henriksen T, Glud AN, Tai Y, Moller Andersen AS, Meier K, Borghammer P, Moro E, Sorensen JCH, Pavese N. Spinal cord stimulation therapy for patients with Parkinson's disease and gait problems (STEP-PD): study protocol for an exploratory, double-blind, randomised, placebo-controlled feasibility trial. BMJ Neurol Open. 2022 Aug 24;4(2):e000333. doi: 10.1136/bmjno-2022-000333. eCollection 2022. PMID 36101543